CLINICAL TRIAL: NCT04415125
Title: Association Between Previous Injury History and Performance of Male Elite Ice Hockey Players
Brief Title: Previous Injury History and Performance of Male Elite Ice Hockey Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, Pt, PhD, Associate Professor, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: University
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Wounds and Injuries; Sports Physical Therapy
Keywords: hockey; performance testing; muscular strength and endurance; wounds and injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- elite male ice hockey players (Experimental): The subjects were 50 elite men's ice hockey players playing in the super league from Turkish clubs subject to Turkey Ice Hockey Federation. All ice hockey players had practicing training programs after warming up for 10 minutes for at least 3 days a week and 1 hour in a day during the season. They also played a match at least 1 day a week. The inclusion criteria were; being a member of Turkish Ice Hockey Federation and to be subject to any of the licensed athletes who played in the super league team, to be over 18, to be male. Exclusion criteria were; being under the age of 18, being a woman, having not suffered a musculoskeletal injury that would prevent him from going to training in the last 1 year or affect the outcome of the measurements.
  Interventions: Diagnostic Test: Applying on-ice and off-ice performance tests

INTERVENTIONS:
Diagnostic Test: Applying on-ice and off-ice performance tests — The subjects were given a written description of study procedures and potential risks.The athletes'history of injury including previous injury site, type, number, date, surgical status, time to return to the field after the injury and the mechanism of injury were recorded. The subjects completed off-ice performance measures followed by on-ice testing with time allotted for warm-up before both the off-ice and on-ice testing.

SUMMARY:
BACKGROUND: In ice hockey, skating is a combination of speed, power, and balance. OBJECTIVE:The aim of this study is to examine the relationship between previous injury history and on-ice and off-ice performance of elite male ice hockey players.

METHODS: This study was designed as prospective cross-sectional study. Fifty elite men's ice hokey players included (n=50, mean age 23y 8mo, SD 5y 3mo). Off-ice performance measures were 30 m Sprint Test, Broad Jump Test, Push-up Test, Hexagon Agility Test, Plank Test. The 2 on-ice tests were 30m On-ice Sprint Test and Cornering "S" Turn Agility Test.The athletes' history of injury were including previous injury site, type, number and the mechanism of injury. RESULTS: In push up test, there was a significant difference in those who had left hand and right knee injuries and, athletes who had dislocation were found to be statistically significant (p <0.05). According to cornering s turn agility test results, athletes who had puck injury were found to be statistically significant (p <0.05). In 30m sprint and hexagon agility test results, athletes who had overuse injury were found to be statistically significant (p <0.05). There was a significant correlation between on-ice 30m sprint and cornering s turn agility tests with broad jump test and also with off-ice push-up and plank tests (p<0.05). CONCLUSIONS: As a result of the performance tests, push up test might be a distinctive test in determining the performance of the athletes after injury. Also on-ice tests had a correlation with off-ice plank test which is the indicator of core muscle strength.

DETAILED DESCRIPTION:
We believe that the current performance and performance deficiencies of the athletes determined and existing training programs will be arranged to eliminate performance deficiencies. We wanted to raise awareness about whether there is a general deficiency in ice hockey performance caused by past injuries and which exercises should be included in the training program in order to overcome performance deficiencies.

ELIGIBILITY:
Inclusion Criteria:

* Being a member of Turkish Ice Hockey Federation,
* To be subject to any of the licensed athletes who played in the super league team
* To be over 18,
* To be male.

Exclusion Criteria:

* Being under the age of 18,
* Being a woman,
* Having not suffered a musculoskeletal injury that would prevent him from going to training in the last 1 year or affect the outcome of the measurements.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
30 meter Sprint Test | 10-15 seconds
  The aim of 30 meter sprint test is to determine acceleration and speed performance of the players
Broad Jump Test | 5-10 seconds
  Lower body muscular power was assessed using Broad Jump Test
Push-up Test | 5-10 minutes
  Upper body strength and muscular endurance were examined by asking each player to complete the maximum number of push-ups
Hexagon Agility Test | 1 minute
  For the hexagon agility test, an equilateral hexagonal with 60 cm on each side was drawn to the ground, the athletes stood in the hexagonand started bouncing off the 6 sides in sequence and jumped back to their original positions. The athletes were reminded that their direction should always be the same when bouncing.The time was started with the start command. The test was stopped at moment he jumped from the last edge into the hexagon
Plank Test | 60 seconds
  Basic plank test was used to evaluate core muscle function of the players
30 meters On-ice Sprint Test | 5-10 seconds
  Sprint ability was evaluated using a simple straight-line sprint test
Cornering "S" Turn Agility Test | 5-10 seconds
  For the Cornering S Turn Agility Test, participants started behind the goal line and net and skated around the two near faceoff circles an S-type fashion

SECONDARY OUTCOMES:
The athletes'history of injury | 5-10 minutes
  The athletes'history of injury including previous injury site, type, number, date, surgical status, time to return to the field after the injury and the mechanism of injury were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Çöük Balcı, Pt,PhD, Study Chair — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)